CLINICAL TRIAL: NCT04765735
Title: Electrically Evoked Compound Action Potentials Human Observation Medtronic Algorithm Comparison Study (ECHO-MAC)
Brief Title: Electrically Evoked Compound Action Potentials Human Observation Medtronic Algorithm Comparison Study
Acronym: ECHO-MAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MDT19024
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Open-loop (OL) testing, then Closed-loop (CL) testing (Experimental): Subjects receive Open-loop testing, then Closed-loop testing (Spinal Cord Stimulation - SCS Therapy)
  Interventions: Device: Open-loop testing, Closed-loop testing - External Spinal Cord Stimulator (SCS)
- Closed-loop testing, then Open-loop testing (Experimental): Subjects receive Closed-loop testing, then Open-loop testing (Spinal Cord Stimulation - SCS Therapy)
  Interventions: Device: Open-loop testing, Closed-loop testing - External Spinal Cord Stimulator (SCS)

INTERVENTIONS:
Device: Open-loop testing, Closed-loop testing - External Spinal Cord Stimulator (SCS) — SCS therapy with an external neurostimulator using either open-loop or closed loop algorithm

SUMMARY:
This is a prospective, multi-center, randomized, single-blind, cross-over, non-significant risk IDE research study to evaluate the in-clinic performance of a closed-loop algorithm in Spinal Cord Stimulation (SCS) therapy with an ENS device.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* Candidate for or undergoing Medtronic SCS device trial for labeled indication - Candidate for or undergoing a Medtronic SCS device trial for labeled indication means that a clinical decision has already been made between a physician and the patient to undergo Medtronic SCS trialing to treat the patient's chronic pain. This decision is to be made prior to discussing with the patient whether to enroll in the study
* Willing and able to provide signed and dated informed consent
* Capable of comprehending and consenting in English
* Willing and able to comply with all study procedures and visits
* Clear, measurable ECAP ECAPs - If during set up of the in-clinic testing, the subject does not have a clear, measurable ECAP (>10uV amplitude obtained consistently and repeatably) they will not move forward with testing or randomization and will be considered a screen failure.

Exclusion Criteria:

* Implanted electrical cardiac devices (e.g., pacemaker, defibrillator)
* Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results (co-enrollment in an interventional study is only allowed when documented pre-approval is obtained from the Medtronic study manager or designee)
* Pregnant or is of child-bearing potential and unwilling to use a medically acceptable form of birth control during the study
* Has untreated major psychiatric comorbidity, as determined by the investigator or designee
* Trialed with a permanent implant lead and extension ("buried lead trial")
* If subject is classified as vulnerable or requires a legally authorized representative (LAR)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Coastal Pain and Spinal Diagnostics, Carlsbad, California
  - Lakewalk Surgery Center, Duluth, Minnesota
  - Nura Research Institute, Edina, Minnesota
  - Twin Cities Pain Clinic, Edina, Minnesota
  - The Ohio State University, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Premier Pain Treatment Institute, Mount Orab, Ohio
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - Innovative Pain Center, Watertown, South Dakota

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized at the In-Clinic Testing Visit following their Enrollment/Baseline Visit (consent visit). Ten Subjects exited the study prior to randomization resulting in 42 subjects that were randomized.
Groups:
- Open-loop Testing, Then Closed-loop Testing: Subjects receive Open-loop testing, then Closed-loop testing (Spinal Cord Stimulation - SCS Therapy)
  Open-loop testing, Closed-loop testing - External Spinal Cord Stimulator (SCS): SCS therapy with an external neurostimulator using either open-loop or closed loop algorithm
Period: Overall Study
Arm/Group | Open-loop Testing, Then Closed-loop Testing | Closed-loop Testing, Then Open-loop Testing
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intent-to-treat (ITT) Analysis Set: Includes all subjects who were randomized.
Arm/Group | Intent-to-treat (ITT) Analysis Set
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5
  Not Reported | 1
  White | 35
  American Indian or Alaska Native | 1
Region of Enrollment [Number; unit: participants]
  United States | 42
Primary Indication for SCS [Count of Participants; unit: Participants]
  Complex Regional Pain Syndrome | 0
  Degenerative Disk Disease | 9
  Failed Back Surgery Syndrome | 3
  Multiple Back Operations | 0
  Postlaminectomy Pain | 17
  Radicular Pain Syndrome | 13

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With a Reduction in Overstimulation Sensation With SCS Using a Closed-loop Algorithm Compared With SCS in Open-loop
Description: For every overstimulation sensation brought about by protocol-prescribed activities, subjects will rate the intensity of the sensation using a 5-point Likert scale. The average intensity score during OL and CL periods will be calculated for each subject. If the average intensity score during CL period is less than that from the OL period, the subject is considered as a subject with a reduction in overstimulation sensation during CL vs. OL period. The primary endpoint is the proportion of subjects with a reduction in overstimulation sensation among subjects who have in-clinic testing.
Time Frame: In-clinic testing (1 day)
Population: Intent-to-treat analysis set included all subjects who were randomized. Analysis was pre-specified in the study statistical analysis plan to report out on the total proportion of subjects with success together, regardless of the randomization sequence.
Measure: Count of Participants; unit: Participants
Groups:
- Intent-to-treat (ITT): Includes all subjects who were randomized.
Arm/Group | Intent-to-treat (ITT)
Number analyzed (Participants) | 42
Participants | 41
Statistical Analysis 1: Comparison: Intent-to-treat (ITT); Test type: Superiority; p < 0.001, Binomial Exact Test — It is hypothesized that the proportion of subjects with a reduction in overstimulation sensation during CL compared to OL period exceeds a performance goal of 50%. H0: p ≤ 50% HA: p > 50%

ADVERSE EVENTS:
Time Frame: The extent of exposure in this study was defined as the time from in-clinic testing to subject discontinuation, which included the exposure to both the OL and CL in-clinic testing. The extent of exposure for all subjects was within 1 day.
Description: Adverse events related to the ECHO-MDT system were collected during the study based on the investigator's assessment of the relationship to the ECHO-MDT system, procedure, or therapy.
Arm/Group | Intent-to-treat (ITT)
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the Clinical Investigation Plan: All proposed publications must be reviewed and approved by Medtronic prior to publication. If required by a publisher, the principal investigator agrees to obtain all necessary authorizations from study subjects prior to submitting study-related information for publication.

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT04765735/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT04765735/SAP_001.pdf